CLINICAL TRIAL: NCT07179055
Title: An Eight-Week, Double-Masked, Randomized, Placebo-Controlled, Phase 2, Evaluation of the Safety and Efficacy of VSJ-110 Ophthalmic Solution in the Treatment of Dry Eye
Brief Title: An Eight-Week Study to Evaluate the Safety and Efficacy of VSJ-110 Compared to Placebo in the Treatment of Dry Eye
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VSJ-110-2202
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- VSJ-110 Solution (Experimental)
  Interventions: Drug: VSJ-110
- Placebo Solution (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSJ-110 — ophthalmic solution
  Arms: VSJ-110 Solution
Drug: Placebo — ophthalmic solution
  Arms: Placebo Solution

SUMMARY:
The purpose of this study is to determine the safety and efficacy of VSJ-110 compared to placebo in the treatment of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age of either gender and any race.
* Provide written informed consent and sign the HIPAA form.
* Be willing and able to follow all instructions and attend all study visits.

Exclusion Criteria:

* Use of any of the disallowed medications during the washout and study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Corneal Staining | Measured over an 8-week treatment period
  Corneal Staining will be assessed by the investigator on a scale of 0-4, with a higher number indicating a higher grade of staining.

SECONDARY OUTCOMES:
Schirmer's Tear Test | Measured over an 8-week treatment period
  Schirmer tear test strips are used to measure ocular fluid.
Eye Dryness Score (EDS) of the Visual Analogue Scale (VAS) | Measured over an 8-week treatment period
  EDS is reported by the subject using a 100-point scale (0=no discomfort and 100=maximum discomfort).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Vanda Investigational Site, Newport Beach, California
  - Vanda Investigational Site, Andover, Massachusetts
  - Vanda Investigational Site, Shelby, North Carolina
  - Vanda Investigational Site, Memphis, Tennessee
  - Vanda Investigational Site, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No